CLINICAL TRIAL: NCT01383031
Title: Randomized Controlled Trial Of Transumbilical Laparoendoscopic Single Site Cholecystectomy Versus Conventional Laparoscopic Cholecystectomy
Brief Title: Safety and Efficacy Study of Transumbilical Laparoendoscopic Single Site Cholecystectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Beijing Friendship Hospital, Beijing Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFH-007
Record Dates: First submitted 2011-06-17; First posted 2011-06-28 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2010-10

CONDITIONS: Gallstone; Gallbladder Polyps
Keywords: laparoscopic cholecystectomy; single site; randomized controlled trail
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Cholecystectomy (Active Comparator): Laparoscopic cholecystectomy（4 ports or 3 ports）will be performed in a routine fashion by one full time faculty member with fellowship training in laparoscopy.
  Interventions: Procedure: CLC
- TU-LESSC (Active Comparator): TU-LESSC will be performed in a routine fashion which is same to CLC（conventional laparoscopic cholecystetomy）by one full time faculty member with fellowship training in laparoscopy through the conventional laparoscopic instruments.
  Interventions: Procedure: TU-LESSC

INTERVENTIONS:
Procedure: CLC — CLC（4 ports or 3 ports）will be performed in a routine fashion by one full time faculty member with fellowship training in laparoscopy.
  Other Names: conventional laparoscopic cholecystectomy
  Arms: Laparoscopic Cholecystectomy
Procedure: TU-LESSC — TU-LESSC will be performed in a routine fashion which is same to CLC by one full time faculty member with fellowship training in laparoscopy through the conventional laparoscopic instruments.
  Other Names: Transumbilical laparoendoscopic single site cholecystectomy
  Arms: TU-LESSC

SUMMARY:
The purpose of this study is to scientifically evaluate the safety, efficacy and cosmetic results of transumbilical laparoendoscopic single site cholecystectomy.

DETAILED DESCRIPTION:
As the natural orifice during embryonic, the transumbilical surgery not only can mask the abdominal scar and avoid infection produced by puncturing stomach, vagina or rectum in NOTES,but also can be played by the conventional laparoscopic instruments. TU-LESS (transumbilical laparoendoscopic single site surgery), is considered to be the most feasible NOTES(natural orifice transluminal endoscopic surgery)technology at present. Researches about TU-LESS mostly are case reports and small samples or the control experiments up to now,there are not persuasive randomized controlled trail between TU-LESS and conventional laparoscopic cholecystectomy. So the investigators design this prospective randomized controlled trail to scientifically evaluate the safety, efficacy and cosmetic results of transumbilical laparoendoscopic single site cholecystectomy .

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 5 Years
* Benign gallbladder diseases
* KPS ≥ 70
* informed consent

Exclusion Criteria:

* Obstructive jaundice
* Broadening of the common bile duct
* Gallstone pancreatitis
* Serious heart,brain,lung, metabolic diseases history
* History of upper abdominal surgery
* Pregnancy or breast-feeding women
* Refuse TU-LESSC
* BMI(Body Mass Index)≥ 30

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
the incidence of surgical complications | up to 12 weeks
  The primary outcome messures are the incidence of surgical complications caused by the two surgeries.Bleeding,bile duct injury and bile leakage during operation.Wound infection，umbilical hernia，poke holes hernia and biliary fistula after operation.

SECONDARY OUTCOMES:
transfer rate | participants will be followed for the duration of hospital stay, an expected average of 5 days
  TU-LESSC（transumbilical laparoendoscopic single site cholecystectomy）is converted to LC（laparoscopic cholecystectomy）or open sugery;LC is converted to open sugery.
quality of life scores | up to 12 weeks
  Count patients' quality of life scores before sugery and at several time points after operation.
pain scores | up to 12 weeks
  Use VAS（Visual Analogue Score）to count patients' pain scores at several time points after operation.
length of hospital stay | participants will be followed for the duration of hospital stay, an expected average of 5 days
total cost of hospitalization | participants will be followed for the duration of hospital stay, an expected average of 5 days
Cosmetic results | 1 month
  Through the incision length and patients' satisfaction to assess cosmetic results.
The incidence of adverse events | up to 12 weeks
  The adverse events occurred after surgery，regardless of whether they are caused by the tow operations。 Such as nausea, dizziness, urinary retention, vomiting and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, doctor, Study Chair — Beijing Friendship Hospital
Locations (1):
- Bejing Friendship Hospital, Beijing, Bejing, China